CLINICAL TRIAL: NCT01170364
Title: Studying the Effects of Sibutramine on Eating Behavior
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to sibutramine being withdrawn from the market.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 5821
Record Dates: First submitted 2010-04-26; First posted 2010-07-27 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: Obesity; sibutramine; eating behavior
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — sibutramine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sibutramine (Experimental): Participants in this arm receive sibutramine 15mg for one week followed by two weeks of placebo.
  Interventions: Drug: Sibutramine; Drug: Placebo
- Placebo (Experimental): Participants are prescribed two weeks of placebo, followed by one week of 15mg sibutramine.
  Interventions: Drug: Sibutramine; Drug: Placebo

INTERVENTIONS:
Drug: Sibutramine — 1 week of active sibutramine (15mg)
  Other Names: Meridia
Drug: Placebo — 2 weeks of placebo
  Other Names: sugar pill

SUMMARY:
Obesity is a major public health concern, and the search for useful pharmacologic interventions is ongoing. This study aims to develop a comprehensive series of assessments to directly assess eating behavior, cognitive functioning, and psychological functioning under sibutramine and placebo conditions.

DETAILED DESCRIPTION:
We will recruit 48 moderately obese men and women seeking weight-loss treatment to participate in a 3-week, randomized, double-blind, cross-over trial of sibutramine 15mg or placebo daily. At the end of weeks 1 and 3, subjects will be asked to participate in a two-day/three-night stay in the Residential Laboratory or Biological Studies Unit of the New York State Psychiatric Institute for comprehensive assessments. The major outcome variable will be the difference in total daily caloric intake between sibutramine and placebo.

Assessments will concentrate on three main components of eating behavior: eating patterns, psychological processing, and neurocognitive function. Eating behavior studies will examine objective variables such as meal size, meal frequency, and subjective aspects of eating such as hunger and fullness. Psychological studies will measure hedonics, including craving, behavioral restraint, and impulsivity. Neurocognitive function assessment will gather information about decision-making, such as the effects of distractors (food and non-food) on task performance. Additionally, drawing from the field of behavioral neuroeconomics, tasks that assess decision-making and the influence of irrational factors on decisions will be assessed. Neuroimaging (fMRI) procedures will also be conducted, and will augment the psychological and neurocognitive assessments by providing a window into the underlying neural circuitry involved.

Following the double-blind phase, participants will be offered open treatment with sibutramine for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* moderately obese
* stable weight for a minimum of 3 months
* systolic blood pressure less than or equal to 140 mm Hg
* diastolic blood pressure less than or equal to 90 mm Hg
* pulse less than or equal to 95 beats per minute
* English language proficiency

Exclusion Criteria:

* on medications known to affect appetite, weight, or metabolism
* current or past history of: binge eating disorder, anorexia nervosa or bulimia nervosa, major depression
* current or past evidence of psychosis, bipolar illness
* current or past history of alcohol or drug abuse or dependence
* known history of learning disorder or developmental disability
* current or past attention deficit hyperactivity disorders
* low platelet count
* current diabetes mellitus
* uncontrolled asthma, or controlled only with oral steroids
* hypothyroidism not adequately treated
* pregnancy, planning to become pregnant, or lactation within the previous 6 months
* history of neurological disorder or injury
* history of moderate or severe head injury
* waist circumference greater than 188 cm
* indwelling metallic object, non-removable metal jewelery, medicinal patch or recent metallic ink tattoo
* pacemaker
* metallic implants
* medication patches
* significant claustrophobia
* color blindness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Mayer, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 potential participants were screened for eligibility between February, 2009 and July 2010 at an academic medical center in New York City, NY.
Pre-assignment Details: 14 of 45 patients were randomized. Of those not randomized, 21 did not meet inclusion criteria.
Groups:
- Sibutramine First, Then Placebo: This is a cross over design study. Participants in this arm begin with one week of 15mg sibutramine, followed by two weeks of placebo.
- Placebo First, Then Sibutramine: This is a cross over design study. Participants in this arm begin with two weeks of placebo, followed by one week of 15mg of sibutramine
Period: Overall Study
Arm/Group | Sibutramine First, Then Placebo | Placebo First, Then Sibutramine
Started | 8 | 6
Completed | 4 | 5 (One participant was unable to begin the second testing period due to scheduling conflicts.)
Not Completed | 4 | 1
Not completed — Protocol Violation | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sibutramine First, Then Placebo: Participants in this group were randomized to begin with 7 days of 15mg of sibutramine, followed by 14 days of placebo.
- Placebo First, Then Sibutramine: Participants in this group were randomized to begin with 14 days of placebo, followed by 7 days of 15mg of sibutramine.
- Total: Total of all reporting groups
Arm/Group | Sibutramine First, Then Placebo | Placebo First, Then Sibutramine | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6) | 39 (11) | 36 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Measured Caloric Intake
Description: The primary outcome measure is 24-hour food intake assessed by 24 hour weighed intake after one week of sibutramine administration compared to one week of placebo administration.
Time Frame: 1 week
Population: This is a cross over design study. All participants received sibutramine and placebo. The sibutramine arm listed here includes all participants who received sibutramine (regardless of whether they received it first or second). The placebo arm included all those who received placebo (regardless of whether they received it first or second).
Measure: Mean (Standard Deviation); unit: kcal
Groups:
- Sibutramine: In this arm, participants received sibutramine 15mg for 7 days
- Placebo: In this arm, participants received placebo (for 15mg sibumtramine) for 7 days.
Arm/Group | Sibutramine | Placebo
Number analyzed (Participants) | 9 | 9
kcal | 1923 (655) | 2373 (774)
Statistical Analysis 1: Comparison: Sibutramine vs Placebo; Test type: Superiority; p < 0.004, paired sample t-test, two tailed

ADVERSE EVENTS:
Time Frame: One week for each intervention.
Description: At assessment visits, participants were asked about the presence or absence of 22 common medication side effects.
Groups:
- Sibutramine: Participants who received sibutramine 15mg capsule every morning for 7 days.
- Placebo: Participants who received a placebo capsule (matching sibutramine 15mg) every morning for 7 days.
Arm/Group | Sibutramine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 7/9 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sibutramine (N=9) | Placebo (N=9)
headache (Nervous system disorders) | 2 | 1
constipation (Gastrointestinal disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 0 | 1
increased appetite (Gastrointestinal disorders) | 0 | 2
difficulty sitting still (Nervous system disorders) | 1 | 0
irregular heartbeat (Cardiac disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0
dry mouth (Gastrointestinal disorders) | 2 | 0
decreased appetite (Gastrointestinal disorders) | 7 | 2
tremor or shakiness (Nervous system disorders) | 1 | 0
sour taste (General disorders) | 1 | 0
trouble sleeping (Nervous system disorders) | 2 | 1
nervousness (Psychiatric disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Early termination of the study given the withdrawal of sibutramine from the US market.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No